CLINICAL TRIAL: NCT04256265
Title: An Expanded Access Program for Risdiplam in Patients With Type 1 or Type 2 Spinal Muscular Atrophy
Brief Title: An Expanded Access Program for Risdiplam in Participants With Spinal Muscular Atrophy (SMA)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AL41887
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam

INTERVENTIONS:
Drug: Risdiplam — Risdiplam will be administered orally once daily

SUMMARY:
This expanded access program (EAP) will provide access to risdiplam for eligible participants with Type 1 or Type 2 spinal muscular atrophy (SMA) before it is commercially available in the United States for the indication of SMA.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Not eligible for treatment with currently approved treatments for SMA, or cannot continue treatment with currently approved medications as documented by the treating physician, or in the treating physician's judgment, the participant is at risk of lack/loss of treatment efficacy of the current therapy.
* The participant does not qualify for and has no access to SMA treatment in the context of an ongoing clinical trial.
* Adequately recovered from any acute illness at the time of screening, and considered clinically well enough to participate, in the opinion of the treating physician.
* Participants with retinopathy of prematurity should have evidence of stable disease.

Type 1 SMA Participants:

- Confirmed diagnosis of 5q-autosomal recessive SMA.

Type 2 SMA Participants:

* Confirmed diagnosis of 5q-autosomal recessive SMA.
* Negative blood pregnancy test at screening (all women of childbearing potential, including those who have had a tubal ligation), and agreement to comply with measures to prevent pregnancy and restrictions on egg and sperm donation.
* Males with female partners of reproductive potential must agree to use highly effective contraception during therapy, and for at least 4 months after treatment discontinuation.

Exclusion Criteria:

* Inability to meet program requirements.
* Concomitant or previous participation in any investigational drug or device study within 90 days prior to screening or 5 half-lives, whichever is longer.
* Administration of other SMN-2 targeting therapy within 120 days of starting risdiplam therapy.
* Administration of SMA gene therapy within the last 3 months (12 weeks) of receiving risdiplam therapy.
* Any serious medical condition, treatment, or abnormality in clinical laboratory tests that, in the treating physician's judgment, precludes the participant's safe participation in the program.
* Ascertained or presumptive hypersensitivity (e.g., anaphylactic reaction) to risdiplam or to the constituents of its formulation.
* Suspicion of illicit drug or alcohol abuse, in the treating physician's judgment.
* Any prior use of an inhibitor or inducer of flavin-containing monooxygenases 1 (FMO1) or flavin-containing monooxygenases 3 (FMO3) taken within 2 weeks (or within 5 times the elimination half-life, whichever is longer) prior to dosing.

Min Age: 2 Months | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (29):
- United States (29):
  - Arkansas Children's Hospital; Pediatrics, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado in Denver-Anschutz Medical Campus, Aurora, Colorado
  - Nemours Children's Hospital, Orlando, Florida
  - Comprehensive NeuroBehavioral Institute, Plantation, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Ann and Robert H. Lurie Children Hospital of Chicago, Chicago, Illinois
  - Southern Illinois University, School of Medicine, Springfield, Illinois
  - Indiana Hemophilia & Thrombosis center, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Massachusetts General Hospital; Neurology, Boston, Massachusetts
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - University of Mississippi Medical Center; Neurology, Jackson, Michigan
  - Gillette Spcl Children's Clin; Pediatric Endocrinology, Saint Paul, Minnesota
  - St. Louis Children Hospital, St Louis, Missouri
  - Goryeb Children's Hospital, Morristown, New Jersey
  - Northwell Hospital, New Hyde Park, New York
  - NYU Langone, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Akron Childrens Hospital, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Virginia Children's Hospital; Developmental, Charlottesville, Virginia
  - University of Wisconsin American Family; Childrens Hospital, Madison, Wisconsin
  - Childrens Hospital of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin

REFERENCES:
- [Derived] Kwon JM, Arya K, Kuntz N, Phan HC, Sieburg C, Swoboda KJ, Veerapandiyan A, Assman B, Bader-Weder S, Dickendesher TL, Hansen J, Lin H, Yan Y, Rao VK; US Expanded Access Program Working Group. An expanded access program of risdiplam for patients with Type 1 or 2 spinal muscular atrophy. Ann Clin Transl Neurol. 2022 Jun;9(6):810-818. doi: 10.1002/acn3.51560. Epub 2022 May 14. PMID 35567422